CLINICAL TRIAL: NCT00372450
Title: A Quality of Life Comparison in Patients With Malignant Dysphagia Treated With Either Self-Expanding Plastic Stents (SEPS) or Self-Expanding Metal Stents (SEMS)
Brief Title: Plastic Stents Compared With Metal Stents in Treating Patients With Malignant Dysphagia Caused by Esophageal Cancer or Gastroesophageal Junction Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: J05109; CDR0000489157 (Registry Identifier: PDQ (Physician Data Query)); JHOC-J05109; NA_00001547 (Other: JHM IRB)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2008-11

CONDITIONS: Esophageal Cancer; Gastrointestinal Complications
Keywords: recurrent esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus; gastrointestinal complications
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus

INTERVENTIONS:
Procedure: management of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Placing a stent in the esophagus may lessen swallowing difficulties and improve quality of life in patients with malignant dysphagia caused by esophageal cancer or gastroesophageal junction cancer.

PURPOSE: This randomized clinical trial is studying self-expanding plastic stents to see how well they work compared with self-expanding metal stents in treating patients with malignant dysphagia caused by esophageal cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess differences from baseline in health-related quality of life of patients with malignant dysphagia due to cancer of the esophagus or gastroesophageal junction palliated with self-expanding plastic stents (SEPS) compared to those who receive self-expanding metal stents (SEMS).

Secondary

* Perform a cost-effective analysis of each type of stent by independent evaluation of the rates of SEPS-related and SEMS-related morbidity that necessitates repeat endoscopic interventions and/or additional healthcare costs in these patients.
* Analyze effective palliation (degree and duration of improvement of dysphagia) in these patients.
* Determine the individual rates of complication associated with each type of esophageal stent in these patients.

OUTLINE: This is a randomized, controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo placement of a self-expanding metal stent on day 1.
* Arm II: Patients undergo placement of a self-expanding plastic stent on day 1. Health-related quality of life is assessed at baseline, 30 days, and 3 months.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary cancer of the esophagus or gastroesophageal junction

  * Squamous cell or other type
* Diagnosis of malignant dysphagia
* Disease deemed surgically inoperable, but may be any of the following:

  * Locally contained
  * Locally advanced
  * Metastatic
  * Unresponsive to previous chemoradiotherapy
  * Recurrent despite previous surgical resection
* Must be either an inpatient OR outpatient at Johns Hopkins Hospital
* No known tracheal compression by tumor burden

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Life expectancy ≥ 6 months
* Platelet count > 50,000/mm³
* INR < 1.5

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior surgery, chemotherapy, biologic therapy, or radiotherapy allowed
* No concurrent surgery, chemotherapy, biologic therapy, or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Estimated); Primary Completion 2008-04-11 (Actual); Study Completion 2008-04-11 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life from baseline to 30 days and 3 months after self-expanding plastic stent or self-expanding metal stent placement

SECONDARY OUTCOMES:
Cost effectiveness of each type of stent
Degree and duration of improvement of dysphagia
Stent-related morbidities
Time to event (time until first complication)
Overall rate of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Jagannath, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States